CLINICAL TRIAL: NCT01121445
Title: The Impact of Daily Sinus Irrigation on Nasal Symptoms in Continuous Positive Airway Pressure (CPAP) Users - A Pilot Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bridgeport Hospital (Other)
Collaborators: NeilMed Pharmaceuticals (Industry)
Responsible Party: Jeff Kwon, MD/Associate Director of Sleep Medicine, Bridgeport Hospital Department of Medicine
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: IRB #041001
Record Dates: First submitted 2010-05-06; First posted 2010-05-12 (Estimated); Last update posted 2010-05-12 (Estimated); Status verified 2010-05

CONDITIONS: Obstructive Sleep Apnea
Keywords: Sleep apnea; CPAP; Saline irrigation
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea Syndromes

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- CPAP with heated humidification (No Intervention): Standard of care
  Interventions: Device: NeilMed nose and sinus irrigation

INTERVENTIONS:
Device: NeilMed nose and sinus irrigation — Saline irrigation used daily plus CPAP with heated humidification for 4 weeks

SUMMARY:
Continuous positive airway pressure (CPAP) is the most commonly used treatment for obstructive sleep apnea. Nasal symptoms such as dryness, itching and congestion are common in CPAP users. Nasal and sinus saline irrigation has been shown to improve these symptoms in individuals with chronic nasal congestion and sinusitis. This is an 8 week study that investigates whether daily saline nasal and sinus irrigation reduces nasal symptoms in patients using CPAP, improves quality of life and CPAP compliance.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Apnea/hypopnea index ≥ 10
* A documented successful CPAP titration

Exclusion Criteria:

* Conditions that in the judgment of the investigator would interfere with subject participation in the study
* History of sinus or nasal surgery
* History of psychiatric illness
* Use of sleep aids, sedatives or narcotics
* Use of oral of subcutaneous anti-coagulants (i.e. warfarin, enoxaparin)
* Bilevel or other nocturnal ventilation other than CPAP
* Use of supplemental oxygen
* Pregnancy or lactating
* Inability or unwillingness to provide informed consent
* Inability to perform baseline measurements
* Inability to be contacted by phone

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2010-05; Primary Completion 2011-03 (Estimated); Study Completion 2011-03 (Estimated)

PRIMARY OUTCOMES:
RQLQ (Rhinoconjunctivitis Quality of Life Questionnaire) | 4 weeks
  A 28-item, self administered questionnaire measuring nasal symptoms and other domains, including activity limitations and eye symptoms. Subjects will be asked to rate their symptoms on a 7-point scale (0=no impairment, 6=severely impaired). Change in RQLQ with daily saline irrigation in CPAP users is the primary outcome of interest.

SECONDARY OUTCOMES:
Epworth Sleepiness Scale | 4 weeks
  The Epworth Sleepiness Scale is a self administered questionnaire that measures subjective daytime hypersomnia on a scale of 0 to 24.
SF-36 | 4 weeks
  The Medical Outcome Study 36-Item Short Form health survey (SF-36) is a 36-item questionnaire which measures 8 domains of health: physical functioning, physical problems, emotional problems, social functioning, mental health, energy/vitality, pain, and general perception of health status. This questionnaire has been used as a validated measure of change in the quality of life of OSA patients on CPAP therapy.
CPAP compliance | 4 weeks
  CPAP card compliance data will be measured to determine if use of daily sinus rinse is associated with an increase in CPAP use. The % of days CPAP used over 4 weeks and the average number of hours of CPAP use per night are the outcomes of interest.

CONTACTS AND LOCATIONS:
Overall Officials: Jeff S Kwon, MD, Principal Investigator — Bridgeport Hospital
Locations (1):
- Bridgeport Hospital, Bridgeport, Connecticut, United States